CLINICAL TRIAL: NCT00281645
Title: A Multicenter Standard of Care-Controlled Study to Evaluate the Long-Term Safety of Bicifadine for the Treatment of Chronic Low Back Pain
Brief Title: Long-Term Safety Study of Bicifadine for the Treatment of Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DOV Pharmaceutical, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOV-075-022
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Last update posted 2007-03-27 (Estimated); Status verified 2007-03

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — bicifadine; Standard of Care

INTERVENTIONS:
Drug: Bicifadine
Drug: Standard of Care (pharmacological analgesic treatment)

SUMMARY:
The primary objective of the study is to evaluate the safety and efficacy of bicifadine 400 mg BID for up to one year in patients with moderate to severe chronic low back pain.

The secondary objectives are to compare the long-term safety of bicifadine to standard of care therapy, to evaluate the safety of bicifadine following discontinuation of dosing, and to evaluate the safety and efficacy of lower doses of bicifadine in patients who do not tolerate bicifadine 400 mg BID.

DETAILED DESCRIPTION:
There are two ways by which subjects could enter this study.

Subjects who completed 12 weeks of treatment in two other double blind clinical studies of bicifadine (Studies 020 and 021, both in the United States) could roll over into this study.

Also, de novo subjects (that is, subjects who had not previously received bicifadine) could enroll in this study.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with low back pain assessed as Class 1, Class 2 or Class 3 according to the Quebec Task Force Classification for Spinal Disorders and without detectable leg weakness on neurological examination.
* Patients must have required on average daily analgesics for the treatment of low back pain over the past 3 months prior to screening.

Main Exclusion Criteria:

* Patients may not have moderate or severe pain in a location other than the lower back (with the exception of radiation to the lower extremity) or weakness in the lower extremities.
* Patients must not have had epidural corticosteroid injections in the lower back within 1 month prior to baseline.
* Patients may not have an unstable medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250
Dates: Start 2004-12

PRIMARY OUTCOMES:
Adverse Events
Clinical Labs
Vital Signs
ECGs

SECONDARY OUTCOMES:
Pain Severity Rating (VAS)
Short-Form McGill Pain Questionnaire (SF-MPQ)
Roland-Morris Disability Questionnaire (RDQ)
Short-Form 36 (SF-36) Health Survey
Patient Withdrawal Checklist